CLINICAL TRIAL: NCT06887140
Title: Prognostic Value of Right Ventricular-pulmonary Arterial Coupling Assessed by Echocardiography in Septic Patients: A Prospective Observational Study
Brief Title: Prognostic Value of Right Ventricular-pulmonary Arterial Coupling Assessed by Echocardiography in Septic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 173/GCN-HDDD
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: Sepsis; Septic shock; Sepsis-induced Cardiomyopathy; Right ventricle-pulmonary artery coupling; Echocardiography
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic patients not having right ventricle-pulmonary artery uncoupling
  Interventions: Diagnostic Test: Echocardiography
- Septic patients having right ventricle-pulmonary artery uncoupling
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — * First echocardiography: within 24 hours after study enrollment,
  * Second echocardiography: 48-72 hours after the initial echocardiography.
  * The recorded echocardiographic parameters include:
    * Morphological and Functional Parameters
    * Mitral Valve Flow Parameters
    * Tissue Doppler Echocardiography Parameters
    * STE Parameters for Left Ventricle Assessment
    * STE Parameters for Right Ventricle Assessment

SUMMARY:
Sepsis and septic shock are common clinical conditions, representing a significant healthcare challenge due to their high mortality rates and increasing incidence. Sepsis-induced cardiomyopathy is a frequent complication, occurring in up to 44% of septic patients. This condition is associated with a two- to three-fold increase in mortality. Although sepsis-induced cardiomyopathy is typically diagnosed via echocardiography to assess left ventricular systolic function, both ventricles may be affected. Several studies have demonstrated that right ventricular dysfunction (RVD)/ right ventricular failure (RVF) was prevalent in sepsis and septic shock, with significant implications for prognosis and mortality.

The right ventricle (RV) has a distinct anatomical structure and function compared to the left ventricle, characterized by its high sensitivity to afterload variations. Even minor increases in afterload can severely impair RV contractile function. Meanwhile, septic patients often experience hypoxemic respiratory failure and require mechanical ventilation. This condition generates hypoxia-induced pulmonary vasoconstriction, which, combined with positive pressure ventilation, leads to increased pulmonary vascular resistance and elevated pulmonary arterial pressure. Additionally, systemic vasodilation reduces RV preload, while septic shock and vasopressor use further compromise right coronary perfusion, exacerbating RV contractile dysfunction. Consequently, simultaneous assessment of RV contractility and its afterload is crucial in septic patients.

Tricuspid annular plane systolic excursion (TAPSE) is a widely used echocardiographic parameter for evaluating RV systolic function. Pulmonary artery systolic pressure (sPAP) reflects RV afterload and can be estimated in the presence of tricuspid regurgitation. Recently, the TAPSE/sPAP ratio has been proposed as a clinical tool to assess right ventricle-pulmonary artery (RV-PA) coupling. This index has been shown to be associated with mortality in patients with pulmonary hypertension and heart failure. Several studies have been conducted to evaluate RV-PA coupling in sepsis and septic shocks, but these studies have limitations in terms of study design and patient selection.

In Vietnam, the issues of RVD/RVF in sepsis/septic shock have not been thoroughly investigated. Le Minh Khoi and colleagues reported that the incidence of reduced RV strain in septic patients was as high as 55.1%. Currently, no studies have specifically evaluated RV function, nor have any studies assessed RV-PA coupling in septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sepsis,
* Received treatment in the Intensive Care Unit (ICU) at the University Medical Center at Ho Chi Minh City during the study period.

Exclusion Criteria:

* Pregnancy,
* History of right ventricular myocardial infarction,
* Acute coronary syndrome within the past 1 week,
* Valvular heart diseases or a history of valve replacement surgery,
* Congenital heart diseases or conditions involving intracardiac shunts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients received treatment in the Intensive Care Unit (ICU) at the University Medical Center at Ho Chi Minh City during the study period
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Feb 2027

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Feb 2027
Length of stay in Intensive Care Unit | Feb 2027
Length of stay in hospital | Feb 2027
Mortality in Intensive Care Unit | Feb 2027

CONTACTS AND LOCATIONS:
Overall Officials: Khoi M Le, A/Prof. Dr., Study Chair — University Medical Center Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Ehrman RR, Sullivan AN, Favot MJ, Sherwin RL, Reynolds CA, Abidov A, Levy PD. Pathophysiology, echocardiographic evaluation, biomarker findings, and prognostic implications of septic cardiomyopathy: a review of the literature. Crit Care. 2018 May 4;22(1):112. doi: 10.1186/s13054-018-2043-8. PMID 29724231
- [Background] Konstam MA, Kiernan MS, Bernstein D, Bozkurt B, Jacob M, Kapur NK, Kociol RD, Lewis EF, Mehra MR, Pagani FD, Raval AN, Ward C; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; and Council on Cardiovascular Surgery and Anesthesia. Evaluation and Management of Right-Sided Heart Failure: A Scientific Statement From the American Heart Association. Circulation. 2018 May 15;137(20):e578-e622. doi: 10.1161/CIR.0000000000000560. Epub 2018 Apr 12. PMID 29650544
- [Background] Mikkelsen ME, Shah CV, Meyer NJ, Gaieski DF, Lyon S, Miltiades AN, Goyal M, Fuchs BD, Bellamy SL, Christie JD. The epidemiology of acute respiratory distress syndrome in patients presenting to the emergency department with severe sepsis. Shock. 2013 Nov;40(5):375-81. doi: 10.1097/SHK.0b013e3182a64682. PMID 23903852
- [Background] Wang S, Bashir Z, Chen EW, Kadiyala V, Sherrod CF, Has P, Song C, Ventetuolo CE, Simmons J, Haines P. Invasive Mechanical Ventilation Is Associated with Worse Right Ventricular Strain in Acute Respiratory Failure Patients. J Cardiovasc Dev Dis. 2024 Aug 9;11(8):246. doi: 10.3390/jcdd11080246. PMID 39195154
- [Background] Repesse X, Charron C, Vieillard-Baron A. Acute respiratory distress syndrome: the heart side of the moon. Curr Opin Crit Care. 2016 Feb;22(1):38-44. doi: 10.1097/MCC.0000000000000267. PMID 26627538
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Guazzi M, Naeije R. Pulmonary Hypertension in Heart Failure: Pathophysiology, Pathobiology, and Emerging Clinical Perspectives. J Am Coll Cardiol. 2017 Apr 4;69(13):1718-1734. doi: 10.1016/j.jacc.2017.01.051. PMID 28359519
- [Background] Jentzer JC, Anavekar NS, Reddy YNV, Murphree DH, Wiley BM, Oh JK, Borlaug BA. Right Ventricular Pulmonary Artery Coupling and Mortality in Cardiac Intensive Care Unit Patients. J Am Heart Assoc. 2021 Apr 6;10(7):e019015. doi: 10.1161/JAHA.120.019015. Epub 2021 Mar 28. PMID 33775107
- [Result] Charpentier J, Luyt CE, Fulla Y, Vinsonneau C, Cariou A, Grabar S, Dhainaut JF, Mira JP, Chiche JD. Brain natriuretic peptide: A marker of myocardial dysfunction and prognosis during severe sepsis. Crit Care Med. 2004 Mar;32(3):660-5. doi: 10.1097/01.ccm.0000114827.93410.d8. PMID 15090944
- [Result] Vallabhajosyula S, Kumar M, Pandompatam G, Sakhuja A, Kashyap R, Kashani K, Gajic O, Geske JB, Jentzer JC. Prognostic impact of isolated right ventricular dysfunction in sepsis and septic shock: an 8-year historical cohort study. Ann Intensive Care. 2017 Sep 7;7(1):94. doi: 10.1186/s13613-017-0319-9. PMID 28884343
- [Result] Vieillard-Baron A, Prigent A, Repesse X, Goudelin M, Prat G, Evrard B, Charron C, Vignon P, Geri G. Right ventricular failure in septic shock: characterization, incidence and impact on fluid responsiveness. Crit Care. 2020 Nov 1;24(1):630. doi: 10.1186/s13054-020-03345-z. PMID 33131508
- [Result] Lanspa MJ, Cirulis MM, Wiley BM, Olsen TD, Wilson EL, Beesley SJ, Brown SM, Hirshberg EL, Grissom CK. Right Ventricular Dysfunction in Early Sepsis and Septic Shock. Chest. 2021 Mar;159(3):1055-1063. doi: 10.1016/j.chest.2020.09.274. Epub 2020 Oct 14. PMID 33068615
- [Result] Guazzi M, Bandera F, Pelissero G, Castelvecchio S, Menicanti L, Ghio S, Temporelli PL, Arena R. Tricuspid annular plane systolic excursion and pulmonary arterial systolic pressure relationship in heart failure: an index of right ventricular contractile function and prognosis. Am J Physiol Heart Circ Physiol. 2013 Nov 1;305(9):H1373-81. doi: 10.1152/ajpheart.00157.2013. Epub 2013 Aug 30. PMID 23997100
- [Result] Zhang H, Lian H, Zhang Q, Chen X, Wang X, Liu D. Prognostic implications of tricuspid annular plane systolic excursion/pulmonary arterial systolic pressure ratio in septic shock patients. Cardiovasc Ultrasound. 2020 Jun 12;18(1):20. doi: 10.1186/s12947-020-00198-y. PMID 32532300
- [Result] Bowcock EM, Gerhardy B, Huang S, Orde S. Right ventricular outflow tract Doppler flow analysis and pulmonary arterial coupling by transthoracic echocardiography in sepsis: a retrospective exploratory study. Crit Care. 2022 Oct 3;26(1):303. doi: 10.1186/s13054-022-04160-4. PMID 36192793
- [Result] Ma Q, Ding C, Wei W, Su C, Li B, Zhou Z, Chen C, Liu B, Zhang X, Wu J. The value of right ventricular pulmonary artery coupling in determining the prognosis of patients with sepsis. Sci Rep. 2024 Jul 3;14(1):15283. doi: 10.1038/s41598-024-65738-2. PMID 38961249
- See also: Le Minh Khoi, Tran Thanh Toan, Dang Hoang Vu, Bui Thi Hanh Duyen, Phan Vu Anh Minh. Feasibility of speckle tracking echocardiographyand myocardial strain impairment in septic patients. Ho Chi Minh City Journal of Medicine. 2021;25(1):56-62. — https://nsti.vista.gov.vn/publication/download/hE/qFPIDsUeZhP.html